CLINICAL TRIAL: NCT01061905
Title: Behavioral Economics Concepts Influencing Healthy Food Choice - Pilot 2
Brief Title: Behavioral Economics and Food Choice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, J. Jane S. Jue, RWJF Clinical Scholar, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: WhartonAramark-BehavEcon-2
Record Dates: First submitted 2010-01-29; First posted 2010-02-03 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Obesity; Overweight
Keywords: health behavior; behavioral economics; calorie labeling; exercise
MeSH Terms: conditions — Obesity; Overweight; Health Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Calorie information only (Experimental): Posting calorie information of sugar-sweetened and zero-calorie beverages prominently on a poster.
  Interventions: Behavioral: Calorie information
- Exercise Equivalent Information (Experimental): Posting of only exercise equivalents (e.g. 45 minutes on a treadmill) for both sugar-sweetened and zero-calorie beverages, prominently on a poster.
  Interventions: Behavioral: Exercise Equivalent only
- Calorie and Exercise Equivalent information (Experimental): Posting of both calorie and exercise equivalent information for both sugar-sweetened and zero-calorie beverages, prominently on a poster.
  Interventions: Behavioral: Calorie & Exercise equivalent information

INTERVENTIONS:
Behavioral: Calorie information — Posting of Calorie information for sugar-sweetened and zero-calorie beverages
  Arms: Calorie information only
Behavioral: Exercise Equivalent only — Posting of only exercise equivalents (e.g. 45 minutes on a treadmill) for both sugar-sweetened and zero-calorie beverages, prominently on a poster.
  Arms: Exercise Equivalent Information
Behavioral: Calorie & Exercise equivalent information — Posting of both calorie and exercise equivalents information for both sugar-sweetened and zero-calorie beverages, prominently on a poster.
  Arms: Calorie and Exercise Equivalent information

SUMMARY:
This is the second in a series of pilot interventions we are conducting to assess how principles from behavioral economics can be applied to improve consumers' food choices. In collaboration with Aramark, the food service vendor, we intend to examine if calorie labeling in different formats impacts consumers choice of bottled beverages in hospital cafeterias. Specifically, we will be testing whether signage that conveys to consumers the number of calories in each bottled beverage will increase the number of zero-calorie beverages sold relative to non-zero-calorie beverages. Likewise, we will test whether signage that conveys calories in exercise equivalents increases the sale of zero-calorie beverages. Lastly, we will test if signage conveying standard calorie information in conjunction with exercise equivalents increases the sale of zero-calorie beverages. We will measure the differential effect of each of these three formats for calorie information.

DETAILED DESCRIPTION:
Individual behavior plays a central role in the disease burden faced by society. Many major health problems in the United States such as obesity are exacerbated by unhealthy behaviors. In our research, we apply ideas from behavioral economics, which integrates concepts from psychology and economics, to the problem of changing health behaviors. In our research we use several of the decision biases that ordinarily lead people to self-harming behavior, to promote healthy behaviors instead. To date, we have been applying this approach to areas such as smoking cessation, weight loss and medication compliance. We were approached by Aramark to collaborate on projects to test the applicability of this approach to changing food choice. Successful pilots in this area would greatly contribute to ongoing discussions nationally on curbing the obesity epidemic. Our plan was to structure interventions to take advantage of the fact that individuals put disproportionate value on present relative to future costs and benefits, known as present-biased preferences. Present-biased preferences can be made to steer people toward healthier options if they are given immediate rewards for healthy behaviors with even small rewards, if they are immediate. Our first project with Aramark used price discounts on zero-calorie beverages as a means to make the benefits of healthier beverage choice more immediate and tangible. At 4 Aramark hospital cafeteria sites, we discounted the price of zero-calorie beverages by 10% and sought to determine the impact on consumers choice of these beverages. At this time, the intervention has just completed, and data analysis is ongoing. Besides financial incentives, as we used in our first pilot project, conveying information can also make the value of future costs and benefits more immediate. It is this principle which we plan to test with the second pilot.

This pilot intervention will use a quasi-experimental, factorial design to test the impact of calorie information presented on posters in different formats on beverage choice (zero-calorie beverage versus other drinks). At each of 4 hospital cafeteria sites, we will conduct 3 separate, consecutive interventions in which we post the following displays for bottled beverages: (A) calorie information, (B) calories plus calories as exercise equivalents, (C) calories as exercise equivalents. Each intervention will last 3 weeks with a 1 week "washout" period (no display) in between interventions. Therefore, the interventions will run for a total of 11 weeks. The order of interventions will be randomized at each site to address ordering effects. Data on bottled beverage sales (zero-calorie vs. non-zero-calorie) will be collected and analyzed at the cafeteria-level. This includes point-of-sale data, inventory, and stock-keeping-units (SKU) data of zero-calorie and regular beverages sold weekly at each site, before, during and after the pilot. In order to make appropriate comparisons across cafeterias, already-conducted site-specific demographic market research analysis on customers (in aggregate) will also be considered. No individual-level consumer data will be collected, obtained, or analyzed in this study.

The unit of analysis for these studies are hospital cafeterias and cafes which are operated by Aramark, the food services company. The cafeterias and cafes are located in a variety of hospitals located nationwide. Through discussions with Aramark, these cafeterias have volunteered to participate in this study. Representatives from Aramark have been in contact with representatives from the hospitals regarding their participation. We expect 4 Aramark sites will participate, which in total will include 6 cafeterias and 3 convenience stores. During the intervention, customers at each site will see the calorie information displays but will be under no obligation to purchase any of the beverages involved in the study.

The 11 week intervention is set to begin in early February. Data on beverage sales at each site will be collected in the weeks and months leading up to the intervention and in the weeks and months following the intervention.

There will be no individual-level data collection, only aggregate monitoring of cafeteria beverage inventory. As such there is almost no risk to human subjects, their privacy, or confidentiality.

Potential risks to humans include altered food choice that negatively affects their health. Though we will be promoting healthier options, there is a very small possibility that such promotion paradoxically may influence individuals to seek out less healthy items. There is also a small risk of such promotions such as exercise labeling to effect individuals psychologically in unexpected ways. The likelihood of both of these is very small and the seriousness of these risks also are minor.

ELIGIBILITY:
Inclusion Criteria:

* Aramark Hospital Cafeteria or Cafe with the ability to provide sales data

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Primary outcome data will comprise of weekly sales and inventory reports provided by each cafeteria. Specifically, we will obtain total sales of the relevant beverages before, during, and after the study. | Weekly sales data collected duing intervention from 2/8/10 through 5/23/10

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD, PhD, Principal Investigator — University of Pennsylvania; J. Jane S. Jue, MD, Principal Investigator — Robert Wood Johnson Foundation Clinical Scholars Program at the University of Pennsylvania; Matthew J Press, MD, Principal Investigator — Robert Wood Johnson Foundation Clinical Scholars Program at the University of Pennsylvania; David Asch, MD, MBA, Principal Investigator — University of Pennsylvania; George Loewenstein, PhD, Principal Investigator — Carnegie Mellon University
Locations (4):
- United States (4):
  - ARAMARK healthcare at North Shore University Health System, Evanston, Illinois
  - ARAMARK Healthcare at Henry Ford Hospital, Detroit, Michigan
  - ARAMARK healthcare at Main Line Health, Bryn Mawr, Pennsylvania
  - ARAMARK healthcare at Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Volpp KG, Pauly MV, Loewenstein G, Bangsberg D. P4P4P: an agenda for research on pay-for-performance for patients. Health Aff (Millwood). 2009 Jan-Feb;28(1):206-14. doi: 10.1377/hlthaff.28.1.206. PMID 19124872
- [Background] Loewenstein G, Brennan T, Volpp KG. Asymmetric paternalism to improve health behaviors. JAMA. 2007 Nov 28;298(20):2415-7. doi: 10.1001/jama.298.20.2415. No abstract available. PMID 18042920
- [Background] Brownell KD, Frieden TR. Ounces of prevention--the public policy case for taxes on sugared beverages. N Engl J Med. 2009 Apr 30;360(18):1805-8. doi: 10.1056/NEJMp0902392. Epub 2009 Apr 8. No abstract available. PMID 19357400
- [Result] Volpp KG, Troxel AB, Pauly MV, Glick HA, Puig A, Asch DA, Galvin R, Zhu J, Wan F, DeGuzman J, Corbett E, Weiner J, Audrain-McGovern J. A randomized, controlled trial of financial incentives for smoking cessation. N Engl J Med. 2009 Feb 12;360(7):699-709. doi: 10.1056/NEJMsa0806819. PMID 19213683
- [Result] Volpp KG, Loewenstein G, Troxel AB, Doshi J, Price M, Laskin M, Kimmel SE. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res. 2008 Dec 23;8:272. doi: 10.1186/1472-6963-8-272. PMID 19102784
- [Result] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Result] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Result] Flegal KM, Graubard BI, Williamson DF, Gail MH. Excess deaths associated with underweight, overweight, and obesity. JAMA. 2005 Apr 20;293(15):1861-7. doi: 10.1001/jama.293.15.1861. PMID 15840860